CLINICAL TRIAL: NCT01386489
Title: VRC 016: A Phase 1b Open-Label, Randomized Clinical Trial to Evaluate Early Innate and Adaptive Immune Responses to the Investigational HIV-1 Vaccines: VRC-HIVADV014-00-VP and VRC-HIVDNA016-00-VP in Ad5 Seronegative Healthy Adults
Brief Title: Immune Responses to Two Experimental HIV Vaccines in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110197; 11-I-0197
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-03-19

CONDITIONS: HIV Negative; Adaptive Immunity; Innate Immunity
Keywords: HIV-uninfected; Mucosal Immunity; Kinetics; Cytokines; Chemokines; Healthy Volunteer; HV

INTERVENTIONS:
Biological: VRC-HIVDNA016-00-VP
Biological: VRC-HIVADV014-00-VP

SUMMARY:
Background:

The primary focus of the Vaccine Research Center (VRC) at the NIH is to develop vaccines for HIV/AIDS. The main purpose of this study is to look in detail at the body s immune response to two experimental HIV vaccines currently in development at the VRC. One is known as the rAd5 vaccine and the other is known as the DNA vaccine. These vaccines are made with pieces of manufactured DNA. They do not contain live or killed HIV. It is impossible for study vaccines to give you HIV and they cannot cause you to give HIV to someone else. Both of these experimental vaccines have been given to people before in other research studies. They have not been approved for treating or preventing HIV infection.

Purpose:

The main purpose of this study is to look in detail at the body s immune responses after the experimental HIV vaccines are given and to assess safety of the study vaccines.

Eligibility:

Healthy volunteers between the ages of 18 and 50 who are not infected with HIV and who meet the eligibility requirements.

Design:

Participants will be screened with a medical history (including questions about sexual history and drug use), physical exam, and blood tests.

The study will have two groups:

<TAB>One group will receive one injection of the rAd5 vaccine, and have 8 clinic visits over 3 months.

<TAB>The second group will have three injections of the DNA vaccine, one injection of the rAd5 vaccine, and have 12 clinic visits over 6 months.

All participants will be asked to provide blood and body fluid samples for testing during the study.

Payment for participation will be provided....

DETAILED DESCRIPTION:
Study Design:

This is a hypothesis-generating descriptive study to evaluate the kinetics and pattern of early innate and adaptive immune responses to the VRC recombinant adenoviral vector serotype 5 vaccine, VRC-HIVADV014-00-VP (rAd5). The rAd5 vaccine has been previously administered to more than 1000 study subjects and characterized as safe and immunogenic. A difference in the pattern of vaccine antigen-specific immune responses observed when rAd5 is given as a single agent compared to after priming by a 6-plasmid DNA vaccine, VRCHIVDNA016-00-VP, has previously been reported. This study will randomize vaccine-naive subjects to receive a single injection of rAd5 or to the DNA primerAd5 boost regimen that is now in a large Phase II study. Collection of blood, rectal, oral and genital specimens for characterization of early innate and adaptive immune responses will follow receipt of rAd5. The hypothesis is that the pattern of early innate and adaptive immune responses elicited by the rAd5 vaccine administered after priming with DNA vaccine will be distinctly different from the pattern elicited when rAd5 is administered as a single agent. The primary objectives are to describe the kinetics and pattern of early innate and adaptive immune responses that occur in blood samples early after administration of rAd5 vaccine alone and after administration following 3 DNA prime injections. Secondary and exploratory objectives are related safety, as well as the pattern of immune responses in mucosal samples and in blood samples.

Product Description:

VRC-HIVDNA016-00-VP [6-plasmid DNA vaccine] is composed of 6 closed, circular DNA plasmids that encode for HIV-1 Gag, Pol and Nef proteins (from clade B) and Env glycoproteins from clade A, clade B, and clade C, which are combined in equal proportions. All injections will be at 4 mg dose in a 1 mL volume administered intramuscularly (IM) by Biojector (registered trademark) into deltoid muscle.

VRC-HIVADV014-00-VP (rAd5 vaccine) is composed of 4 recombinant nonreplicating adenoviral vectors that encode for HIV-1 Gag/Pol polyproteins (from clade B) and Env glycoproteins from clade A, clade B, and clade C, which are combined in a 3:1:1:1 ratio, respectively, in a final formulation buffer (FFB). All injections will be at 10(10) PU dose in a 1 mL volume administered IM by needle and syringe into deltoid muscle.

Subjects:

The study target accrual is at least 20 subjects who complete collection of blood, oral, rectal and genital specimens through 2 weeks after the rAd5 vaccination. To account for potential discontinuations from the study, enrollment may include up to 36 HIV-uninfected adults, ages 18-50 years old that are HIV vaccine-naive and adenovirus serotype 5 (Ad5) antibody negative at screening; males must be fully circumcised.

Study Plan:

Subjects will be randomized at a 1:1 ratio to receive a single injection of rAd5 or the DNA prime-rAd5 boost schedule and will be stratified by gender to achieve approximately equal distribution of each gender into the two vaccination schedules. Subjects randomized to Group 1 may receive the vaccination on enrollment day or schedule the day of vaccination to occur within 6 weeks followed by the expected 24 hours in the inpatient unit and day 3 post-vaccination sample collections for the frequent sampling that will immediately ensue according to the sample collection schedule. Subjects randomized to Group 2 will receive the first of three DNA vaccinations and schedule projected dates for the subsequent injections and timepoints with intensive sample collection schedules. Due to the need to commit to about 3 days of disruption in normal daily activities, starting with the day of rAd5 vaccination on either schedule, flexibility in scheduling of the rAd5 vaccination is included in the protocol plan.

Subjects from both groups will be admitted to the NIH Clinical Center overnight for the first 24 hours following vaccination with rAd5. On the rAd5 vaccination day, peripheral blood samples will be collected for serum, plasma and peripheral blood mononuclear cells at seven target time points in the first 24 hours as follows: pre-injection and post-injection hours 1, 3, 6, 12, 18 and 24; then days 3, 5, 7, 14 and 28 post-rAd5 vaccine. Mucosal sampling will occur on day 14 after rAd5 vaccine. This will include buccal mucosa, rectal secretions, cervical secretions (from women) and semen samples (from men). There will be a blood collection to assess innate immunity following the 3rd DNA vaccination in Group 2 with blood draws at pre-injection and at post-injection hours 1, 3, 6 and 18.

The safety of vaccinations and the research plan will be monitored by a protocol safety review team.

Study Duration:

Subjects will be followed in the clinic through 12 weeks after last study injection and contacted for long term follow-up 12 weeks later and then every 48 weeks through Study Week 144.

ELIGIBILITY:
* INCLUSION CRITERIA:

A volunteer must meet all of the following criteria:

1. 18 to 50 years old.
2. No prior vaccinations with an HIV vaccine or adenoviral vector vaccine.
3. Available for clinical follow-up for up to 36 weeks after enrollment and committed to follow-up contacts through 144 weeks after enrollment.
4. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
5. Able and willing to complete the informed consent process.
6. Willing to donate oral, rectal and genital secretion samples and blood samples for research that will be stored and used for future research.
7. Willing to discuss HIV infection risks with the study clinicians, assessed as low risk for HIV infection, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required clinic visit in the protocol schedule.
8. In good general health without clinically significant medical history.
9. Physical examination and laboratory results without clinically significant findings and a weight 50 kg or more with body mass index (BMI) less than or equal to 40 within the 56 days prior to enrollment.

   Laboratory Criteria within 56 days prior to enrollment:
10. Hemoglobin greater than or equal to 11.2 g/dL for women; greater than or equal to 13.0 g/dL for men.
11. White blood cells (WBC) = 3,000-12,000 cells/mm(3).
12. Differential and platelet count either within institutional normal range or accompanied by site physician approval.
13. Alanine aminotransferase (ALT) less than or equal to 1.75 times upper limit of normal.
14. HIV-uninfected as evidenced by a negative FDA-approved HIV diagnostic blood test or negative HIV polymerase chain reaction (PCR) test.
15. Seronegative (defined as less than 1:12) for adenovirus serotype 5 antibody as measured by the NVITAL assay within 84 days (12 weeks) prior to enrollment.

    Male-Specific Criterion:
16. A male participant must be fully circumcised as assessed by screening physical examination.

    Female-Specific Criteria:
17. Negative Beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.
18. A female participant must meet any of the following pregnancy prevention criteria:

No reproductive potential because of menopause [one year without menses] or because of tubal ligation,

or

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through 12 weeks after the last vaccination on the study schedule,

or

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through 12 weeks after the last vaccination on the study schedule by one of the following methods:

* condoms, male or female, with or without a spermicide
* diaphragm or cervical cap with spermicide
* intrauterine device
* contraceptive pills or patch, vaginal ring, injection or other FDA-approved contraceptive method
* male partner has previously undergone a vasectomy.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

1. Woman who is breast-feeding or planning to become pregnant during study participation.
2. Woman who is known to not have a cervix or who report having a clinically significant abnormal Pap smear without a subsequent normal result.

   Volunteer has received any of the following substances:
3. Systemic immunosuppressive medications or cytotoxic medications within the 12 weeks prior to enrollment. [With the exception that a short course (duration of 10 days or less or a single injection) of corticosteroids for a self-limited condition at least 2 weeks prior to enrollment in the study will not exclude study participation.]
4. Blood products or immunoglobulin within 56 days (8 weeks) prior to enrollment.
5. Investigational research agents within 28 days (4 weeks) prior to enrollment.
6. Live attenuated vaccines within 28 days (4 weeks) prior to enrollment.
7. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days (2 weeks) prior to enrollment.
8. Current anti-tuberculosis prophylaxis or therapy.

   Volunteer has a history of any of the following clinically significant conditions:
9. Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain.
10. Clinically significant autoimmune disease or immunodeficiency.
11. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
12. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
13. Thyroid disease that is not well controlled.
14. A history of hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
15. Generalized idiopathic urticaria within the 1 year prior to enrollment.
16. Hypertension that is not well controlled by medication.
17. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
18. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
19. Seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years.
20. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
21. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; disorder requiring lithium; or within five years prior to enrollment, history of a suicide plan or attempt.
22. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-06-17; Primary Completion 2014-03-09 (Actual); Study Completion 2014-03-19 (Actual)

PRIMARY OUTCOMES:
To describe the kinetics and patterns over the time of innate and adaptive immunologic responses in peripheral blood as well as the pattern of adaptive immune responses at a single timepoint in mucosal samples following vaccination with the rAd5...

SECONDARY OUTCOMES:
To assess the safety and tolerability of the investigational vaccines.

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Ledgerwood, D.O., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] McElrath MJ, Haynes BF. Induction of immunity to human immunodeficiency virus type-1 by vaccination. Immunity. 2010 Oct 29;33(4):542-54. doi: 10.1016/j.immuni.2010.09.011. PMID 21029964
- [Background] Borrow P, Shattock RJ, Vyakarnam A; EUROPRISE Working Group. Innate immunity against HIV: a priority target for HIV prevention research. Retrovirology. 2010 Oct 11;7:84. doi: 10.1186/1742-4690-7-84. PMID 20937128
- [Background] Koup RA, Roederer M, Lamoreaux L, Fischer J, Novik L, Nason MC, Larkin BD, Enama ME, Ledgerwood JE, Bailer RT, Mascola JR, Nabel GJ, Graham BS; VRC 009 Study Team; VRC 010 Study Team. Priming immunization with DNA augments immunogenicity of recombinant adenoviral vectors for both HIV-1 specific antibody and T-cell responses. PLoS One. 2010 Feb 2;5(2):e9015. doi: 10.1371/journal.pone.0009015. PMID 20126394